CLINICAL TRIAL: NCT05853601
Title: Theophylline Prophylaxis During Hypothermia to Limit Neonatal Nephron Damage
Acronym: TheoPHyLNNe
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Collaborators: University of Oklahoma (Other)
Responsible Party: Principal Investigator, Jeffrey Segar, Professor, Department of Pediatrics, Medical College of Wisconsin
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: PRO46949
Record Dates: First submitted 2023-03-20; First posted 2023-05-11 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-03

CONDITIONS: Acute Kidney Injury; HIE
MeSH Terms: conditions — Acute Kidney Injury | interventions — Theophylline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Single Dose Theophylline (Experimental): Single dose of theophylline or aminophylline (5mg/kg IV) given within 18 hours after birth
  Interventions: Drug: Single Dose Theophylline
- Repeat Dose Theophylline (Experimental): Loading dose of theophylline or aminophylline (5mg/kg IV) given within 18 hours of birth, with two subsequent doses (1.2 mg/kg IV) given at 12 and 24 hours after the loading dose
  Interventions: Drug: Repeat Dose Theophylline
- Standard treatment (No Intervention): Infants cared for according to standard practice.

INTERVENTIONS:
Drug: Single Dose Theophylline — Subjects are given a single loading dose of theophylline, 5mg/kg IV, within 18 hours after birth. A bioequivalent dose of aminophylline, a more soluble, ethylenediamine salt of theophylline, may be substituted for theophylline. The bioequivalent dose of aminophylline is 120% of the theophylline dose.
  Arms: Single Dose Theophylline
Drug: Repeat Dose Theophylline — Subjects are given a loading dose of theophylline, 5mg/kg IV, within 18 hours of birth, and then two subsequent doses (1.2mg/kg iv) at 12 hours and 24 hours after loading dose. A bioequivalent dose of aminophylline, a more soluble, ethylenediamine salt of theophylline, may be substituted for theophylline. The bioequivalent dose of aminophylline is 120% of the theophylline dose.
  Arms: Repeat Dose Theophylline

SUMMARY:
Acute kidney injury is a significant complication for infants who experience hypoxic ischemic encephalopathy, being associated with increased rates of death and prolonged hospitalization. This pilot study of theophylline administration soon after birth for the prevention of kidney injury will lay the foundation for the conduct of a larger clinical trial that seeks to identify a theophylline as a novel therapy to prevent kidney injury in thousands of at-risk infants.

DETAILED DESCRIPTION:
Acute kidney injury (AKI) is commonly seen in infants diagnosed with hypoxic-ischemic encephalopathy (HIE) and is associated with increased rates of morbidity and mortality. Currently, there are no approved therapies that target the prevention of AKI. Several small trials in infants with HIE suggest that a single dose of theophylline given soon after birth attenuates the development of AKI. However, these studies were not performed in infants being treated with therapeutic hypothermia (the current standard of care for moderate to severe HIE), and only reported short-term outcomes. Therefore, few clinicians use theophylline in the management of these patients. The long-term goal is to undertake an appropriately powered multicenter clinical trial to test the hypothesis that for infants > 35 weeks gestation treated with therapeutic hypothermia for HIE, intravenous theophylline (or aminophylline) within the first 18 hours after birth will result in a decreased incidence and/or severity of AKI or death (composite primary outcome) and improved long-term (2 year) renal outcomes. Before the conduct of a large trial, the feasibility of implementing the intervention and ability to measure relevant clinical outcomes need to be demonstrated. Therefore, the investigators propose a small pilot and feasibility clinical trial to i) evaluate recruitment, protocol adherence, and data collection procedures in a therapeutic trial of theophylline to decrease the incidence of AKI or death compared to standard treatment in infants with HIE being treated with therapeutic hypothermia; ii) evaluate the utility and applicability of established measures (serum creatinine, urine output, fluid balance) and novel, exploratory approaches to identify AKI in infants; and iii) determine theophylline pharmacokinetic, pharmacodynamic, safety and preliminary effectiveness profiles of two different theophylline dosing regimens in a therapeutic trial of theophylline to decrease the incidence of AKI or death compared to standard treatment. Using a mixed methods data analysis strategy to assess the research and intervention process and examine outcomes of the intervention, the investigators will generate the requisite data to inform development and implementation of an appropriately powered study to determine whether theophylline attenuates the risk and severity of AKI in infants with HIE treated with therapeutic hypothermia.

ELIGIBILITY:
Inclusion Criteria:

* gestational age at birth >= 35 weeks by best obstetrical dating
* birth weight > 1800 grams
* clinical determination of HIE and treatment with hypothermia being initiated within six hours of birth according to institutional guidelines
* no known congenital abnormalities involving the brain, kidneys, heart or lungs
* ability to administer theophylline via intravenous route within 18 hours of birth

Exclusion Criteria:

* infants with suspected or diagnosed significant renal, urinary tract, brain, heart, or lung abnormalities
* infant with known chromosomal anomaly
* evidence of head trauma or skull fracture causing major intracranial hemorrhage
* inability to initiate hypothermia within six hours of birth
* attending physician unwilling to have infant participate in the study
* inability to obtain informed consent within 18 hours of birth

Ages: 1 Hour to 18 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2023-10-17 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
Recruitment of patients | 2 years
  Examine the ability to recruit and enroll patients in trial. We will assess the number of eligible patients and compare that number to those actually enrolled. This ratio will inform regarding the ability to recruit patients in a larger, randomized, appropriately powered trial.

SECONDARY OUTCOMES:
Pharmacokinetic Profile of Theophylline#1 | 2 years
  Evaluate plasma concentrations (mg/dl) of theophylline at time points ranging from 30 minutes to 48 hours after dosing
Safety profile of theophylline#1 | 2 years
  Incidence of tachycardia (heart rate > 200 beats per minute for 15 minutes) after theophylline dosing defined by pediatric neurologist
Safety profile of theophylline#2 | 2 years
  Incidence of hyperglycemia, defined as two sequential serum glucose values over 200 mg/dl) over one hour apart after theophylline dosing
Safety profile of theophylline#3 | 2 years
  Incidence of clinical seizures as diagnosed by a trained pediatric neurologist
Demonstration of successful adherence to study protocol | 2 years
  Evaluate the incidence of protocol deviations both per subject and study-wide. Incidence will be expressed as number of study violations per enrolled subject
Successful data collection procedures | 2 years
  Percent of incomplete data entry points per subject will be evaluated by reviewing data in REDCap
Successful biospecimen collection procedures | 2 years
  Rate of successful collection and analysis of biospecimens per study logs. Data will be determined as percentage of successful completions (successful completions divided by opportunities per protocol).
Pharmacokinetic Profile of Theophylline#2 | 2 years
  Determine area under the curve profile of serum theophylline concentration (mg/dl) over time (hours) up to 48 hours after dosing of theophylline
Acute kidney injury#1 | 2 years
  Incidence of acute kidney injury as defined by modified neonatal KDIGO criteria using serum creatinine values
Acute kidney injury#2 | 2 years
  Incidence of acute kidney injury as defined by modified neonatal KDIGO criteria using urine output values (ml/kg/hour)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Segar, MD, Principal Investigator — Medical College of Wisconsin
Locations (1):
- University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] DeFronzo R, Fleming GA, Chen K, Bicsak TA. Metformin-associated lactic acidosis: Current perspectives on causes and risk. Metabolism. 2016 Feb;65(2):20-9. doi: 10.1016/j.metabol.2015.10.014. Epub 2015 Oct 9. PMID 26773926
- [Background] Le Tourneau C, Lee JJ, Siu LL. Dose escalation methods in phase I cancer clinical trials. J Natl Cancer Inst. 2009 May 20;101(10):708-20. doi: 10.1093/jnci/djp079. Epub 2009 May 12. PMID 19436029
- [Background] See KC. Metformin-associated lactic acidosis: A mini review of pathophysiology, diagnosis and management in critically ill patients. World J Diabetes. 2024 Jun 15;15(6):1178-1186. doi: 10.4239/wjd.v15.i6.1178. PMID 38983827
- [Background] Liao S, Li D, Hui Z, McLachlan CS, Zhang Y. Metformin added to bosentan therapy in patients with pulmonary arterial hypertension associated with congenital heart defects: a pilot study. ERJ Open Res. 2018 Aug 22;4(3):00060-2018. doi: 10.1183/23120541.00060-2018. eCollection 2018 Jul. PMID 30151369
- [Background] Brittain EL, Niswender K, Agrawal V, Chen X, Fan R, Pugh ME, Rice TW, Robbins IM, Song H, Thompson C, Ye F, Yu C, Zhu H, West J, Newman JH, Hemnes AR. Mechanistic Phase II Clinical Trial of Metformin in Pulmonary Arterial Hypertension. J Am Heart Assoc. 2020 Nov 17;9(22):e018349. doi: 10.1161/JAHA.120.018349. Epub 2020 Nov 10. PMID 33167773
- [Background] Biag HMB, Potter LA, Wilkins V, Afzal S, Rosvall A, Salcedo-Arellano MJ, Rajaratnam A, Manzano-Nunez R, Schneider A, Tassone F, Rivera SM, Hagerman RJ. Metformin treatment in young children with fragile X syndrome. Mol Genet Genomic Med. 2019 Nov;7(11):e956. doi: 10.1002/mgg3.956. Epub 2019 Sep 14. PMID 31520524
- [Background] Ayoub R, Ruddy RM, Cox E, Oyefiade A, Derkach D, Laughlin S, Ades-Aron B, Shirzadi Z, Fieremans E, MacIntosh BJ, de Medeiros CB, Skocic J, Bouffet E, Miller FD, Morshead CM, Mabbott DJ. Assessment of cognitive and neural recovery in survivors of pediatric brain tumors in a pilot clinical trial using metformin. Nat Med. 2020 Aug;26(8):1285-1294. doi: 10.1038/s41591-020-0985-2. Epub 2020 Jul 27. PMID 32719487
- [Background] Hutchinson AM, Pais R, Endginton AN, Pilon B, MacDonald JM, MacDonald ME, Lewis T, Offringa M, Kalish BT. Safety and feasibility trial protocol of metformin in infants after perinatal brain injury. BMJ Paediatr Open. 2025 Aug 24;9(1):e002784. doi: 10.1136/bmjpo-2024-002784. PMID 40850908
- [Background] Kirkpatrick EC, Mitchell ME, Thilly WG, Cava J, Tomita-Mitchell A, Gostjeva EV. Use of Metformin in Pulmonary Vein Stenosis after TAPVR Repair. Glob Pediatr Health. 2020 Sep 25;7:2333794X20958924. doi: 10.1177/2333794X20958924. eCollection 2020. No abstract available. PMID 33029553
- [Background] Alemon-Medina R, Altamirano-Bustamante N, Lugo-Goytia G, Garcia-Alvarez R, Rivera-Espinosa L, Torres-Espindola LM, Chavez-Pacheco JL, Juarez-Olguin H, Gomez-Garduno J, Flores-Perez C, Fernandez-Perez PG. Comparative Bioavailability and Pharmacokinetics Between the Solid Form of Metformin vs a Novel Liquid Extemporaneous Formulation in Children. Dose Response. 2021 Sep 27;19(3):15593258211033140. doi: 10.1177/15593258211033140. eCollection 2021 Jul-Sep. PMID 34602916
- [Background] Park SI, Lee H, Oh J, Lim KS, Jang IJ, Kim JA, Jung JH, Yu KS. A fixed-dose combination tablet of gemigliptin and metformin sustained release has comparable pharmacodynamic, pharmacokinetic, and tolerability profiles to separate tablets in healthy subjects. Drug Des Devel Ther. 2015 Feb 4;9:729-36. doi: 10.2147/DDDT.S75980. eCollection 2015. PMID 25678778
- [Background] Kuhlmann I, Noddebo Nyrup A, Bjerregaard Stage T, Hougaard Christensen MM, Korshoj Bergmann T, Damkier P, Nielsen F, Hojlund K, Brosen K. Oral and intravenous pharmacokinetics of metformin with and without oral codeine intake in healthy subjects: A cross-over study. Clin Transl Sci. 2021 Nov;14(6):2408-2419. doi: 10.1111/cts.13107. Epub 2021 Aug 12. PMID 34268884
- [Background] Rana U, Joshi C, Whitney E, Afolayan A, Dowell J, Teng RJ, Konduri GG. Decreased Liver Kinase B1 Expression and Impaired Angiogenesis in a Murine Model of Bronchopulmonary Dysplasia. Am J Respir Cell Mol Biol. 2024 Oct;71(4):481-494. doi: 10.1165/rcmb.2024-0037OC. PMID 38869353
- [Background] Yadav A, Rana U, Michalkiewicz T, Teng RJ, Konduri GG. Decreased AMP-activated protein kinase (AMPK) function and protective effect of metformin in neonatal rat pups exposed to hyperoxia lung injury. Physiol Rep. 2020 Sep;8(18):e14587. doi: 10.14814/phy2.14587. PMID 32959498
- [Background] Hardie DG, Ross FA, Hawley SA. AMPK: a nutrient and energy sensor that maintains energy homeostasis. Nat Rev Mol Cell Biol. 2012 Mar 22;13(4):251-62. doi: 10.1038/nrm3311. PMID 22436748
- [Background] Ratner V, Starkov A, Matsiukevich D, Polin RA, Ten VS. Mitochondrial dysfunction contributes to alveolar developmental arrest in hyperoxia-exposed mice. Am J Respir Cell Mol Biol. 2009 May;40(5):511-8. doi: 10.1165/rcmb.2008-0341RC. Epub 2009 Jan 23. PMID 19168698
- [Background] Higgins RD, Jobe AH, Koso-Thomas M, Bancalari E, Viscardi RM, Hartert TV, Ryan RM, Kallapur SG, Steinhorn RH, Konduri GG, Davis SD, Thebaud B, Clyman RI, Collaco JM, Martin CR, Woods JC, Finer NN, Raju TNK. Bronchopulmonary Dysplasia: Executive Summary of a Workshop. J Pediatr. 2018 Jun;197:300-308. doi: 10.1016/j.jpeds.2018.01.043. Epub 2018 Mar 16. No abstract available. PMID 29551318
- [Background] Abman SH, Bancalari E, Jobe A. The Evolution of Bronchopulmonary Dysplasia after 50 Years. Am J Respir Crit Care Med. 2017 Feb 15;195(4):421-424. doi: 10.1164/rccm.201611-2386ED. No abstract available. PMID 28199157